CLINICAL TRIAL: NCT03215537
Title: Development of Patient Tailored Guideline of Physical Activity for Lung Cancer Survivor After Surgery; to Improve the Symptoms, Complications and Quality of Life
Brief Title: Development of Patient Tailored Guideline of Physical Activity for Lung Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2015-11-025-002
Record Dates: First submitted 2017-07-05; First posted 2017-07-12 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-02

CONDITIONS: Lung Cancer
Keywords: physical activity; cardiopulmonary function; quality of life; Perioperative management; comprehensive intervention; health behavior model
MeSH Terms: conditions — Lung Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- observation (No Intervention): No Intervention
- comprehensive intervention (Active Comparator): preoperative: exercise counseling postoperative : symptoms counseling and pulmonary rehabilitation
  Interventions: Behavioral: comprehensive intervention

INTERVENTIONS:
Behavioral: comprehensive intervention — preoperative and postoperative exercise program
  Arms: comprehensive intervention

SUMMARY:
This study aims to propose a perioperative comprehensive intervention based on health behavior model to improve cardiopulmonary function and quality of life among lung cancer patients following

DETAILED DESCRIPTION:
This study aims to propose a perioperative comprehensive intervention based on health behavior model to improve cardiopulmonary function and quality of life among lung cancer patients following:

1. understanding multi-dimensional factors affecting cardiopulmonary function and quality of life
2. development of multidisciplinary comprehensive intervention
3. evaluation the effects of comprehensive intervention using cluster design

ELIGIBILITY:
Inclusion Criteria:

* lung cancer patients before surgery

Exclusion Criteria:

* Eastern Cooperative Oncology Group Performance Status <1
* Neoadjuvant therapy
* Multiple cancer
* Recurrent lung cancer.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2016-03-02 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2023-12-02 (Estimated)

PRIMARY OUTCOMES:
Changes of cardiopulmonary function | Baseline, 1 month after surgery, 6 months after surgery, 1year after surgery
  six minute walk test

SECONDARY OUTCOMES:
complication | 1 month after surgery, 6 months after surgery, 1year after surgery
  Pneumonia
Changes of pulmonary function | Baseline, 1 month after surgery, 6 months after surgery, 1year after surgery
  forced expiratory volume at one second, forced vital capacity
Changes of physical activity | Baseline, 1 month after surgery, 6 months after surgery, 1year after surgery
  wearable device
Changes of physical fitness | Baseline, 1 month after surgery, 6 months after surgery, 1year after surgery
  muscle strengths
Changes of quality of life | Baseline, 1 month after surgery, 6 months after surgery, 1year after surgery
  quality of life questionnaire
Changes of Fatigue | Baseline, 1 month after surgery, 6 months after surgery, 1year after surgery
  Fatigue questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jae Ill Zo, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Lee J, Kong S, Shin S, Lee G, Kim HK, Shim YM, Cho J, Kang D, Park HY. Wearable Device-Based Intervention for Promoting Patient Physical Activity After Lung Cancer Surgery: A Nonrandomized Clinical Trial. JAMA Netw Open. 2024 Sep 3;7(9):e2434180. doi: 10.1001/jamanetworkopen.2024.34180. PMID 39302678